CLINICAL TRIAL: NCT02367820
Title: A Phase 3 Multicenter, Open-Label, 52-Week Study To Evaluate the Long-Term Safety and Tolerability of NKTR-181 in Subjects With Moderate to Severe Chronic Low Back Pain or Chronic Non-Cancer Pain
Brief Title: Long-Term Safety and Tolerability Study of NKTR-181 in Subjects With Chronic Low Back Pain or Chronic Non-Cancer Pain
Acronym: SUMMIT-LTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-181-08
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain; Chronic Pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NKTR-181 (Experimental): NKTR-181 twice daily (BID) tablets
  Interventions: Drug: NKTR-181 BID tablets

INTERVENTIONS:
Drug: NKTR-181 BID tablets — NKTR-181 tablets 100-600 mg twice daily (BID)

SUMMARY:
The purpose of this 52-week open label study is to determine the long-term safety of a new opioid molecule, NKTR-181, in patients with moderate to severe chronic low back pain or chronic non-cancer pain.

DETAILED DESCRIPTION:
This is an open-label safety and tolerability study in which approximately 600 subjects will receive NKTR-181 for up to 52 weeks. Subjects may include newly enrolled subjects and subjects who have recently completed SUMMIT-07 study.

This study will also investigate the pharmacokinetics of NKTR-181 in patients with chronic low back pain or chronic non-cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female aged 18 to 75 years old
* Clinical diagnosis of moderate to severe, chronic low back or non-cancer pain for at least three months
* Not experiencing adequate pain relief or have failed previous treatment with non-opioid analgesics
* Opioid analgesia is necessary
* Currently taking no less than 10 mg but no more than 60 mg of morphine sulfate equivalents (MSE) per day of opioid analgesics for at least 7 days prior to entry
* Females of child bearing potential must be using a highly effective form of birth control. All subjects must agree to use double-barrier contraception during participation in this study and for at least 2 months after the last dose of the study drug.
* Willing and able to provide informed consent

Exclusion Criteria:

* History of hypersensitivity, intolerance, or allergy to opioids
* Surgical procedures in the last 4 weeks or plans to undergo surgical procedures during the study period
* Untreated moderate to severe sleep apnea
* Chronic migraines as the primary pain condition
* Cancer related pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- United States (56):
  - Investigator Site - Saraland, Saraland, Alabama
  - Investigator Site - Phoenix, Phoenix, Arizona
  - Investigator Site - Tempe, Tempe, Arizona
  - Investigator Site - Little Rock, Little Rock, Arkansas
  - Investigator Site - Stamford, Stamford, Connecticut
  - Investigator Site - Clearwater, Clearwater, Florida
  - Investigator Site - Fort Lauderdale, Fort Lauderdale, Florida
  - Investigator Site - Fort Myers, Fort Myers, Florida
  - Investigator Site - Jacksonville, Jacksonville, Florida
  - Investigator Site - Orlando, Orlando, Florida
  - Investigator Site - Ormond Beach, Ormond Beach, Florida
  - Investigator Site - Plantation, Plantation, Florida
  - Investigator Site - Tampa, Tampa, Florida
  - Investigator Site - West Palm Beach, West Palm Beach, Florida
  - Investigator Site - Atlanta, Atlanta, Georgia
  - Investigator Site - Blue Ridge, Blue Ridge, Georgia
  - Investigator Site - Marietta, Marietta, Georgia
  - Investigator Site - Norcross, Norcross, Georgia
  - Investigator Site - Gurnee, Gurnee, Illinois
  - Investigator Site - West Des Moines, West Des Moines, Iowa
  - Investigator Site - Wichita, Wichita, Kansas
  - Investigator Site - Louisville, Louisville, Kentucky
  - Investigator Site - Bossier, Bossier City, Louisiana
  - Investigator Site - New Orleans, New Orleans, Louisiana
  - Investigator Site - Shreveport, Shreveport, Louisiana
  - Investigator Site - Bay City, Bay City, Michigan
  - Investigator Site - Pinconning, Pinconning, Michigan
  - Investigator Site - Biloxi, Biloxi, Mississippi
  - Investigator Site - Saint Louis 1, St Louis, Missouri
  - Investigator Site - Saint Louis 2, St Louis, Missouri
  - Investigator Site - Omaha, Omaha, Nebraska
  - Investigator Site - Las Vegas 2, Las Vegas, Nevada
  - Investigator Site - Las Vegas 1, Las Vegas, Nevada
  - Investigator Site - Rochester, Rochester, New York
  - Investigator Site - Williamsville, Williamsville, New York
  - Investigator Site - Greensboro, Greensboro, North Carolina
  - Investigator Site - Winston Salem, Winston-Salem, North Carolina
  - Investigator Site - Fargo, Fargo, North Dakota
  - Investigator Site - Beavercreek, Beavercreek, Ohio
  - Investigator Site - Cincinnati 1, Cincinnati, Ohio
  - Investigator Site - Cincinnati 2, Cincinnati, Ohio
  - Investigator Site - Columbus, Columbus, Ohio
  - Investigator Site - Duncansville, Duncansville, Pennsylvania
  - Investigator Site - Jenkintown, Jenkintown, Pennsylvania
  - Investigator Site - Dakota Dunes, Dakota Dunes, South Dakota
  - Investigator Site - Rapid City, Rapid City, South Dakota
  - Investigator Site - Memphis, Memphis, Tennessee
  - Investigator Site - Arlington, Arlington, Texas
  - Investigator Site - Austin, Austin, Texas
  - Investigator Site - Killeen, Killeen, Texas
  - Investigator Site - San Antonio, San Antonio, Texas
  - Investigator Site - Salt Lake City, Salt Lake City, Utah
  - Investigator Site - West Jordan, West Jordan, Utah
  - Investigator Site - Midlothian, Midlothian, Virginia
  - Investigator Site - Norfolk, Norfolk, Virginia
  - Investigator Site - Kenosha, Kenosha, Wisconsin

REFERENCES:
- [Background] Gudin J, Rauck R, Argoff C, Agaiby E, Gimbel J, Katz N, Doberstein SK, Tagliaferri M, Tagliaferri M, Potts J, Wild J, Lu L, Siddhanti S, Hale M, Markman J. Long-term Safety and Tolerability of NKTR-181 in Patients with Moderate to Severe Chronic Low Back Pain or Chronic Noncancer Pain: A Phase 3 Multicenter, Open-Label, 52-Week Study (SUMMIT-08 LTS). Pain Med. 2020 Nov 7;21(7):1347-1356. doi: 10.1093/pm/pnz169. PMID 31361019
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject screened 14 April 2015. Last subject out: 24 January 2018. The study was conducted at 55 medical/research centers in the United States.
Pre-assignment Details: The titration phase of the study was designed to titrate patients to a dose of NKTR-181 that provided adequate analgesia and acceptable side effects.
Groups:
- NKTR-181: NKTR-181 tablets at 100-600 mg orally twice daily
Period: Overall Study
Arm/Group | NKTR-181
Started | 638
Completed | 402
Not Completed | 236

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set is defined as all enrolled subjects who received at least 1 dose of study drug.
Groups:
- Rollover NKTR-181: Subjects administered NKTR-181 in preceding phase 3 efficacy/safety study
- Rollover PBO: Subjects administered placebo in preceding phase 3 efficacy/safety study
- De Novo Naive: Newly enrolled opioid naïve subjects
- De Novo Opioid Experienced: Newly enrolled opioid experienced subjects
- Total: Total of all reporting groups
Arm/Group | Rollover NKTR-181 | Rollover PBO | De Novo Naive | De Novo Opioid Experienced | Total
Number analyzed (Participants) | 214 | 217 | 73 | 134 | 638
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (12.01) | 51.4 (12.31) | 51.9 (10.44) | 55.6 (11.12) | 52.4 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 126 | 44 | 82 | 375
  Male | 91 | 91 | 29 | 52 | 263
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 0 | 1 | 6
  Asian | 2 | 2 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 71 | 70 | 19 | 24 | 184
  White | 136 | 138 | 51 | 106 | 431
  More than one race | 0 | 1 | 1 | 1 | 3
  Unknown or Not Reported | 2 | 3 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events
Description: Count of subjects reporting treatment emergent adverse events
Time Frame: Screening baseline through end of study, an average of 57 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover NKTR-181 | Rollover PBO | De Novo Opioid Experienced | De Novo Naive
Number analyzed (Participants) | 214 | 217 | 134 | 73
Participants | 138 | 151 | 110 | 62

2. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Pain Intensity Item to Week 52
Description: A self-reported scale measuring severity of pain on function. The mean of the 4 intensity items (3-6) is calculated and used as a measure of pain severity. If there were missing items when the pain severity score was calculated, the mean of the completed items in one dimension (dimensions include pain severity and pain interference) were imputed to substitute the missing item, provided that more than 50% of the items in one dimension were completed (Halling, 1999). The range of pain intensity and interference for each question is from 0 to 10. The range of possible scores is from 0 to 70. Higher score indicates relatively worse pain severity and greater interference that pain causes in day to day activities.
Time Frame: Baseline, monthly change from baseline till the end of study
Population: Safety Analysis Set is defined as all enrolled subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rollover NKTR-181 | Rollover PBO | De Novo Opioid Experienced | De Novo Naive
Number analyzed (Participants) | 185 | 188 | 129 | 72
Scores on a scale
  Pain Intensity: Baseline | 3.57 (1.968) | 4.11 (2.112) | 5.91 (1.749) | 6.18 (1.459)
  Pain Intensity: Change from Baseline to Day 1: number analyzed (Participants) | 173 | 177 | 100 | 52
  Pain Intensity: Change from Baseline to Day 1 | -1.22 (2.109) | -1.71 (2.212) | -2.19 (2.009) | -2.66 (1.808)
  Pain Intensity: Change from Baseline to Day 30: number analyzed (Participants) | 169 | 168 | 92 | 46
  Pain Intensity: Change from Baseline to Day 30 | -1.02 (2.233) | -1.40 (2.314) | -2.26 (2.134) | -2.26 (2.068)
  Pain Intensity: Change from Baseline to Day 60: number analyzed (Participants) | 162 | 161 | 85 | 43
  Pain Intensity: Change from Baseline to Day 60 | -1.28 (2.037) | -1.58 (2.172) | -2.01 (2.000) | -2.49 (1.966)
  Pain Intensity: Change from Baseline to Day 90: number analyzed (Participants) | 149 | 153 | 81 | 41
  Pain Intensity: Change from Baseline to Day 90 | -1.31 (2.142) | -1.48 (2.278) | -2.06 (1.932) | -2.38 (2.115)
  Pain Intensity: Change from Baseline to Day 120: number analyzed (Participants) | 146 | 150 | 75 | 39
  Pain Intensity: Change from Baseline to Day 120 | -1.24 (2.269) | -1.44 (2.267) | -2.04 (1.933) | -2.58 (1.874)
  Pain Intensity: Change from Baseline to Day 150: number analyzed (Participants) | 142 | 146 | 73 | 39
  Pain Intensity: Change from Baseline to Day 150 | -1.28 (2.116) | -1.54 (2.319) | -2.09 (2.016) | -2.44 (2.323)
  Pain Intensity: Change from Baseline to Day 180: number analyzed (Participants) | 143 | 146 | 71 | 37
  Pain Intensity: Change from Baseline to Day 180 | -1.37 (2.103) | -1.49 (2.425) | -1.87 (2.053) | -2.80 (2.173)
  Pain Intensity: Change from Baseline to Day 210: number analyzed (Participants) | 137 | 142 | 68 | 37
  Pain Intensity: Change from Baseline to Day 210 | -1.28 (2.131) | -1.58 (2.220) | -2.06 (1.944) | -3.01 (2.258)
  Pain Intensity: Change from Baseline to Day 240: number analyzed (Participants) | 129 | 133 | 64 | 32
  Pain Intensity: Change from Baseline to Day 240 | -1.15 (1.837) | -1.82 (2.190) | -2.21 (1.908) | -2.84 (2.289)
  Pain Intensity: Change from Baseline to Day 270: number analyzed (Participants) | 120 | 121 | 56 | 31
  Pain Intensity: Change from Baseline to Day 270 | -1.45 (2.154) | -1.62 (2.366) | -1.83 (1.915) | -2.65 (1.933)
  Pain Intensity: Change from Baseline to Day 300: number analyzed (Participants) | 95 | 96 | 39 | 21
  Pain Intensity: Change from Baseline to Day 300 | -1.09 (2.149) | -1.48 (2.303) | -2.08 (2.144) | -2.31 (2.043)
  Pain Intensity: Change from Baseline to Day 364: number analyzed (Participants) | 129 | 129 | 65 | 36
  Pain Intensity: Change from Baseline to Day 364 | -0.78 (2.175) | -1.31 (2.520) | -1.20 (2.102) | -2.15 (2.055)

3. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Pain Interference Item to Week 52
Description: A self-reported scale measuring interference of pain on function. The mean of the 7 interference items was calculated and used as a measure of Pain interference. If there were missing items when the pain interference score was calculated, the mean of the completed items in one dimension (dimensions include pain severity and pain interference) were imputed to substitute the missing item, provided that more than 50% of the items in one dimension were completed (Halling, 1999). The range of pain interference is from 0 to 10. Higher score indicates relatively worse pain problem.
Time Frame: Baseline, monthly change from baseline till the end of study
Population: Safety Analysis Set is defined as all enrolled subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rollover NKTR-181 | Rollover PBO | De Novo Opioid Experienced | De Novo Naive
Number analyzed (Participants) | 185 | 188 | 129 | 72
Scores on a scale
  Pain Interference: Baseline | 2.91 (2.205) | 3.25 (2.281) | 5.41 (2.298) | 5.44 (1.957)
  Pain Interference: Change from Baseline to Day 1: number analyzed (Participants) | 173 | 177 | 100 | 52
  Pain Interference: Change from Baseline to Day 1 | -1.23 (2.301) | -1.52 (2.163) | -2.34 (2.175) | -2.71 (2.169)
  Pain Interference: Change from Baseline to Day 30: number analyzed (Participants) | 169 | 168 | 92 | 46
  Pain Interference: Change from Baseline to Day 30 | -1.07 (2.070) | -1.29 (2.340) | -2.51 (2.583) | -2.17 (2.679)
  Pain Interference: Change from Baseline to Day 60: number analyzed (Participants) | 162 | 161 | 85 | 43
  Pain Interference: Change from Baseline to Day 60 | -1.17 (2.070) | -1.32 (2.104) | -2.18 (2.350) | -2.38 (2.277)
  Pain Interference: Change from Baseline to Day 90: number analyzed (Participants) | 149 | 153 | 81 | 41
  Pain Interference: Change from Baseline to Day 90 | -1.24 (2.344) | -1.34 (2.222) | -2.15 (2.447) | -2.11 (2.179)
  Pain Interference: Change from Baseline to Day 120: number analyzed (Participants) | 146 | 150 | 75 | 39
  Pain Interference: Change from Baseline to Day 120 | -1.31 (2.389) | -1.36 (2.309) | -2.33 (2.299) | -2.48 (2.173)
  Pain Interference: Change from Baseline to Day 150: number analyzed (Participants) | 142 | 146 | 73 | 39
  Pain Interference: Change from Baseline to Day 150 | -1.12 (2.329) | -1.22 (2.500) | -2.26 (2.372) | -2.16 (2.290)
  Pain Interference: Change from Baseline to Day 180: number analyzed (Participants) | 143 | 146 | 71 | 37
  Pain Interference: Change from Baseline to Day 180 | -1.31 (2.247) | -1.33 (2.507) | -2.09 (2.551) | -2.27 (2.404)
  Pain Interference: Change from Baseline to Day 210: number analyzed (Participants) | 137 | 142 | 68 | 37
  Pain Interference: Change from Baseline to Day 210 | -0.95 (2.325) | -1.29 (2.215) | -2.43 (2.365) | -2.38 (2.611)
  Pain Interference: Change from Baseline to Day 240: number analyzed (Participants) | 129 | 133 | 64 | 32
  Pain Interference: Change from Baseline to Day 240 | -0.95 (2.119) | -1.55 (2.197) | -2.49 (2.503) | -2.27 (2.240)
  Pain Interference: Change from Baseline to Day 270: number analyzed (Participants) | 120 | 121 | 56 | 31
  Pain Interference: Change from Baseline to Day 270 | -1.21 (2.339) | -1.37 (2.329) | -2.02 (2.374) | -2.01 (2.193)
  Pain Interference: Change from Baseline to Day 300: number analyzed (Participants) | 95 | 96 | 39 | 21
  Pain Interference: Change from Baseline to Day 300 | -0.90 (2.307) | -1.38 (2.137) | -2.07 (2.280) | -1.94 (2.357)
  Pain Interference: Change from Baseline to Day 364: number analyzed (Participants) | 129 | 129 | 65 | 36
  Pain Interference: Change from Baseline to Day 364 | -0.69 (2.258) | -1.14 (2.493) | -1.33 (2.396) | -2.08 (2.504)

ADVERSE EVENTS:
Time Frame: Adverse events were reported starting immediately after the subject provided written informed consent through the end of study, which was approximately 57-weeks in length for each subject.
Description: Adverse events were collected after the subject provided written informed consent through the end of study. Adverse event data were obtained via spontaneous reports or per direct questioning or observation during protocol-mandated study assessments. All ongoing AEs were followed until resolution or for 14 days after the subject's last visit, whichever came first. All SAEs were followed until resolution, stabilization of condition, return to baseline, or until follow-up was no longer possible.
Arm/Group | Rollover NKTR-181 | Rollover PBO | De Novo Opioid Experienced | De Novo Naive
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/217 | 0/134 | 0/73
Serious Adverse Events (participants affected / at risk) | 10/214 | 8/217 | 8/134 | 4/73
Other Adverse Events (participants affected / at risk) | 136/214 | 151/217 | 110/134 | 62/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover NKTR-181 (N=214) | Rollover PBO (N=217) | De Novo Opioid Experienced (N=134) | De Novo Naive (N=73)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hisoplasmosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover NKTR-181 (N=214) | Rollover PBO (N=217) | De Novo Opioid Experienced (N=134) | De Novo Naive (N=73)
Constipation (Gastrointestinal disorders) | 28 (28) | 41 (41) | 56 (56) | 41 (41)
Nausea (Gastrointestinal disorders) | 17 (17) | 21 (21) | 17 (17) | 21 (21)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 11 (11) | 4 (4) | 8 (8)
Vomiting (Gastrointestinal disorders) | 13 (13) | 10 (10) | 3 (3) | 9 (9)
Drug withdrawal (General disorders) | 10 (10) | 16 (16) | 10 (10) | 2 (2)
Fatigue (General disorders) | 1 (1) | 4 (4) | 4 (4) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 19 (19) | 10 (10) | 7 (7)
Urinary tract infection (Infections and infestations) | 10 (10) | 14 (14) | 5 (5) | 6 (6)
Influenza (Infections and infestations) | 5 (5) | 10 (10) | 4 (4) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7) | 7 (7) | 3 (3)
Headache (Nervous system disorders) | 9 (9) | 21 (21) | 21 (21) | 6 (6)
Somnolence (Nervous system disorders) | 6 (6) | 13 (13) | 9 (9) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3) | 6 (6) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (4) | 5 (5) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a joint manuscript has not been submitted for publication within twelve (12) months of completion or termination of the study, the PI is free to publish separately, upon provision of any proposed publication or manuscript to the Sponsor at least sixty (60) days before it is submitted or otherwise disclosed.

DOCUMENTS (2):
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02367820/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT02367820/SAP_003.pdf